CLINICAL TRIAL: NCT00364793
Title: An Open-label Study of Liquid and Sprinkled Formulations of Efavirenz Administered in Combination With Didanosine and Emtricitabine in HIV-infected Infants and Children 3 Months to 6 Years of Age.
Brief Title: Safety, Tolerability and Pharmacokinetics of Efavirenz in HIV-Infected Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI266-922
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: HIV, Pediatric
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Didanosine; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EFV+ddI+FTC in patients >= 3 months to < 6 months (Experimental): EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle, or oral solution (30 mg/mL. In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and FTC (emtricitabine) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
  Interventions: Drug: Efavirenz (EFV) + Didanosine (ddI) + Emtricitabine (FTC)
- EFV+ddI+FTC in patients >=6 months to < 2 years (Experimental): EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle, or oral solution (30 mg/mL. In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and FTC (emtricitabine) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
  Interventions: Drug: Efavirenz (EFV) + Didanosine (ddI) + Emtricitabine (FTC)
- EFV+ddI+FTC in patients >= 2 years to < 3 years (Experimental): EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle, or oral solution (30 mg/mL. In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and FTC (emtricitabine) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
  Interventions: Drug: Efavirenz (EFV) + Didanosine (ddI) + Emtricitabine (FTC)
- EFV+ddI+FTC in patients >= 3 years to <= 6 years (Experimental): EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle, or oral solution (30 mg/mL. In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and FTC (emtricitabine) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
  Interventions: Drug: Efavirenz (EFV) + Didanosine (ddI) + Emtricitabine (FTC)

INTERVENTIONS:
Drug: Efavirenz (EFV) + Didanosine (ddI) + Emtricitabine (FTC) — Oral Solution, Capsules or Tablets, Oral, once daily
  Efavirenz (EFV) per weight-based dosing nomogram (max 720 mg)
  Didanosine (ddI) 240 mg/m2 (max 400 mg)
  Emtricitabine (FTC) 6 mg/kg (max 200 mg)
  Where EFV oral solution is commercially available: 48 weeks or until 3rd birthday (whichever is longer);
  Where EFV oral solution NOT commercially available: until 7th birthday or until able to swallow EFV capsules (whichever occurs first)
  Other Names: Sustiva; BMS-561525

SUMMARY:
The primary purpose of this study is to find the dose of Efavirenz for young children. The safety and how the medication is tolerated will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected; >=3 months of age to <=6 years of age (at time of treatment); screening plasma viral load >=1000 copies/mL

Exclusion Criteria:

* Genotypic or phenotypic resistance to EFV, ddl, or FTC/lamivudine (3TC) at screening

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2007-02; Primary Completion 2011-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal
- Local Institution, Cali, Colombia
- Mexico (7):
  - Local Institution, Colima, Colima
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Puebla City, Puebla
  - Local Institution, San Luis Potosí City
- Local Institution, Panama City, Panama
- South Africa (3):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Westdene, Gauteng
  - Local Institution, Cape Town, Western Cape
- Local Institution, Bangkok, Thailand

REFERENCES:
- [Derived] Pavia-Ruz N, Rossouw M, Saez-Llorens X, Bunupuradah T, Taylor M, Yang R, Sevinsky H, Krystal M, Lataillade M, Seekins D, Biguenet S. Efavirenz Capsule Sprinkle and Liquid Formulations With Didanosine and Emtricitabine in HIV-1-infected Infants and Children 3 Months to 6 Years of Age: Study AI266-922. Pediatr Infect Dis J. 2015 Dec;34(12):1355-60. doi: 10.1097/INF.0000000000000913. PMID 26379163
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study initiated February 2007 and completed July 2013. All participants enrolled in countries where efavirenz (EFV) oral solution was not commercially available could remain on study until their 7th birthday or until they were able to swallow EFV capsules (whichever occurred first).
Pre-assignment Details: 56 participants were enrolled but 19 were never treated. Reasons for not treating: 2 deaths, 1 lost to follow up, 6 other (not specified), 9 no longer met study criteria, 1 withdrew consent.
Groups:
- EFV+ddI+FTC in Infants >=3 Months to < 6 Months: EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle (eg, yogurt, applesauce, or grape jelly), or oral solution (30 mg/mL); participants unable to meet the desired exposures using the oral solution, or those not able to tolerate the oral solution, used the capsule contents sprinkled on food. In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and emtricitabine (FTC) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
- EFV+ddI+FTC in Infants >=6 Months to < 2 Years; EFV+ddI+FTC in Children >= 2 Years to < 3 Years; EFV+ddI+FTC in Children >= 3 Years to <= 6 Years: EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle (eg, yogurt, applesauce, or grape jelly), or oral solution (30 mg/mL); participants unable to meet the desired exposures using the oral solution, or those not able to tolerate the oral solution, used the capsule contents sprinkled on food. In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and FTC (emtricitabine) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
Period: Overall Study
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Started | 15 | 10 | 4 | 8
Completed | 7 | 5 | 0 | 5
Not Completed | 8 | 5 | 4 | 3
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 3 | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Poor or non-compliance | 1 | 1 | 0 | 1
Not completed — No longer meets criteria | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated participants who received at least one dose of study drug (EFV) were analyzed.
Groups:
- EFV+ddI+FTC in Infants >=3 Months to < 6 Months; EFV+ddI+FTC in Infants >=6 Months to < 2 Years; EFV+ddI+FTC in Children >= 2 Years to < 3 Years; EFV+ddI+FTC in Children >= 3 Years to <= 6 Years: EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle (eg, yogurt, applesauce, or grape jelly), or oral solution (30 mg/mL). In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and FTC (emtricitabine) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
- Total: Total of all reporting groups
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | Total
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
Age, Continuous [Median (Full Range); unit: years] | 0.392 [0.296 to 0.501] | 0.825 [0.586 to 1.906] | 2.313 [2.094 to 2.995] | 3.922 [2.998 to 6.976] | 0.663 [0.296 to 6.976]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 1 | 6 | 13
  Male | 9 | 10 | 3 | 2 | 24
Race/Ethnicity, Customized [Number; unit: participants] — Ethnicity was not collected because the study was conducted outside of the United States.
  participants
    White | 3 | 9 | 4 | 8 | 24
    Black or African American | 7 | 0 | 0 | 0 | 7
    Asian | 2 | 0 | 0 | 0 | 2
    Other | 3 | 1 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Panama | 3 | 0 | 0 | 1 | 4
  Mexico | 2 | 7 | 3 | 7 | 19
  Argentina | 0 | 3 | 1 | 0 | 4
  Thailand | 2 | 0 | 0 | 0 | 2
  South Africa | 7 | 0 | 0 | 0 | 7
  Colombia | 1 | 0 | 0 | 0 | 1
Human Immunodeficiency Virus (HIV) Ribonucleic acid (RNA) Viral Load (log10 c/mL) [Median (Full Range); unit: log10 c/mL] — Human immunodeficiency virus (HIV) ribonucleic acid (RNA) values ≥ 1,000 copies per milliliter (c/mL) were considered evidence of infection. HIV RNA measures the viral load and was first measured using the ultrasensitive and standard Roche Amplicor Polymerase Chain Reaction (PCR), version 1.5, and then the method of measurement was switched to the COBAS AmpliPrep/COBAS TaqMan HIV IVD method.
  log10 c/mL | 5.88 [3.34 to 6.74] | 5.88 [2.12 to 5.88] | 5.88 [4.88 to 5.88] | 5.26 [3.38 to 5.88] | 5.88 [2.12 to 6.74]
HIV RNA Viral Load Category [Number; unit: participants] — Human immunodeficiency virus (HIV) ribonucleic acid (RNA) values greater than, equal to (≥) 1,000 copies per milliliter (c/mL) were considered evidence of infection. Categories listed indicate the plasma viral load prior to study treatment (Baseline). HIV RNA was first measured using the ultrasensitive and standard Roche Amplicor PCR, version 1.5, and then the method of measurement was switched to the COBAS AmpliPrep/COBAS TaqMan HIV IVD method.
  participants
    < 30,000 copies/mL | 3 | 1 | 0 | 1 | 5
    30,000 to <100,000 copies/mL | 0 | 1 | 1 | 2 | 4
    100,000 to <500,000 copies/mL | 2 | 1 | 0 | 2 | 5
    500,000 to <=750,000 copies/mL | 1 | 1 | 0 | 1 | 3
    >750,000 copies/mL | 9 | 6 | 3 | 2 | 20
CD4 Cell Count (n=13, 9, 3, 7, 32) [Median (Full Range); unit: cells/mm^3] — A CD4 cell is an antigenic marker of helper/inducer T cells. These cells were counted during the hematology cell counts performed during a Complete Blood Cell count (CBC) performed by the Central Laboratory. CD4 are measured as number of cells per millimeter to the third power (cells/mm^3). Not all treated participants provided a measurement for this baseline parameter (n=number of participants with this baseline measurement).
  cells/mm^3 | 1785 [200 to 3584] | 1569 [516 to 2879] | 517 [129 to 558] | 540 [11 to 1363] | 1144 [11 to 3584]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) and Plasma Concentration 24 Hours Post-dose (Cmin) of EFV at Week 2 - Pharmacokinetic Evaluable Population
Description: Cmax and Cmin were derived from plasma concentrations versus time using a validated liquid chromatography tandem mass spectrometry method (LC-MS/MS). The lower limit of quantification (LLOQ) for EFV was 10.0 nanograms per milliliter (ng/mL) and the upper limit of quantification (ULOQ) was 8,000 ng/mL. Cmax and Cmin were recorded directly from experimental observations. Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the pharmacokinetic parameters were summarized using geometric means. Cmax and Cmin were measured in ng/mL.
Time Frame: Week 2
Population: All participants who received at least one dose of study drug (EFV) and had adequate pharmacokinetic (PK) profiles were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 3 | 10 | 3 | 7
ng/mL
  Cmax | 3790 (76) | 1998 (51) | 2167 (68) | 2632 (83)
  Cmin | 391 (141) | 445 (57) | 648 (75) | 1185 (111)

2. Secondary Outcome: The Number of Participants With Plasma HIV RNA < 400 Copies Per Milliliter (c/mL) at Week 48 as Analyzed by Different Algorithms - All Treated Participants
Description: Algorithms: Confirmed Virologic Response (CVR) non-completer = failure (NC = F): participants were responders if they achieved confirmed HIV RNA < 400 c/mL at Week 48; participants were failures if virologic rebound occurred at or before Week 48; therapy discontinued before Week 48; no response by Week 48, or missing HIV RNA at Week 48 and beyond. Virologic Response - Observed Cases (VR-OC): participants were responders according to a single on-treatment HIV RNA < 400 c/mL closest to the planned Week 48 visit and within the predefined Week 48 visit window; those on treatment and missing their Week 48 measurement were responders only if previous and subsequent measurements to the Week 48 visit window were < 400 c/mL; denominator was all who remained on treatment through Week 48. Snapshot: participants were responders according to the last on-treatment HIV RNA < 400 c/mL in the predefined Week 48 visit window; denominator was all treated participants.
Time Frame: Week 48
Population: Treated participants, who received at least 1 dose of study drug (EFV), were analyzed. n=number of participants with available on-treatment data for analysis by each algorithm.
Measure: Number; unit: participants
Groups:
- Total Participants: All participants across all age groups, ie greater than, equal to 3 months to less than, equal to 6 years.
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | Total Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  CVR (NC=F) n=15, 10, 4, 8, 37 | 7 | 6 | 3 | 5 | 21
  VR-OC n=9, 9, 3, 6, 27 | 7 | 6 | 3 | 5 | 21
  SNAPSHOT n=15, 10, 4, 8, 37 | 7 | 6 | 3 | 5 | 21

3. Secondary Outcome: The Number of Participants With Plasma HIV RNA Levels < 50 c/mL at Week 48 as Analyzed by Different Algorithms - All Treated Participants
Description: Algorithms: Confirmed Virologic Response (CVR) non-completer = failure (NC = F): participants were responders if they achieved confirmed HIV RNA < 50 c/mL at Week 48; participants were failures if virologic rebound occurred at or before Week 48; therapy discontinued before Week 48; no response by Week 48, or missing HIV RNA at Week 48 and beyond. Virologic Response - Observed Cases (VR-OC): participants were responders according to a single on-treatment HIV RNA < 50 c/mL closest to the planned Week 48 visit and within the predefined Week 48 visit window; those on treatment and missing their Week 48 measurement were responders only if previous and subsequent measurements to the Week 48 visit window were < 50 c/mL; denominator was all who remained on treatment through Week 48. Snapshot: participants were responders according to the last on-treatment HIV RNA < 50 c/mL in the predefined Week 48 visit window; denominator was all treated participants.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- EFV+ddI+FTC in All Participants: All participants across all age groups, ie greater than, equal to 3 months to less than, equal to 6 years who received study drug. EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle (eg, yogurt, applesauce, or grape jelly), or oral solution (30 mg/mL). In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and FTC (emtricitabine) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  CVR (NC=F) n=15, 10, 4, 8, 37 | 6 | 6 | 2 | 4 | 18
  VR-OC n=9, 9, 3, 6, 27 | 6 | 5 | 2 | 4 | 17
  SNAPSHOT n=15, 10, 4, 8, 37 | 6 | 5 | 2 | 4 | 17

4. Secondary Outcome: The Number of Participants With Plasma HIV RNA Levels < 400 c/mL at Week 24 as Analyzed by Different Algorithms - All Treated Participants
Description: Algorithms: Confirmed Virologic Response (CVR) non-completer = failure (NC = F): participants were responders if they achieved confirmed HIV RNA < 400 c/mL at Week 24; participants were failures if virologic rebound occurred at or before Week 24; therapy discontinued before Week 24; no response by Week 24, or missing HIV RNA at Week 24 and beyond. Virologic Response - Observed Cases (VR-OC): participants were responders according to a single on-treatment HIV RNA < 400 c/mL closest to the planned Week 24 visit and within the predefined Week 24 visit window; those on treatment and missing their Week 24 measurement were responders only if previous and subsequent measurements to the Week 24 visit window were < 400 c/mL; denominator was all who remained on treatment through Week 24.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  CVR (n=15, 10, 4, 8, 37) | 8 | 7 | 4 | 7 | 26
  VR-OC(n=11,10 ,4, 7, 32) | 8 | 7 | 4 | 6 | 25

5. Secondary Outcome: The Number of Participants With Plasma HIV RNA Levels < 50 c/mL at Week 24 as Analyzed by Different Algorithms - All Treated Participants
Description: Algorithms: Confirmed Virologic Response (CVR) non-completer = failure (NC = F): participants were responders if they achieved confirmed HIV RNA < 50 c/mL at Week 24; participants were failures if virologic rebound occurred at or before Week 24; therapy discontinued before Week 24; no response by Week 24, or missing HIV RNA at Week 24 and beyond. Virologic Response - Observed Cases (VR-OC): participants were responders according to a single on-treatment HIV RNA < 50 c/mL closest to the planned Week 24 visit and within the predefined Week 24 visit window; those on treatment and missing their Week 24 measurement were responders only if previous and subsequent measurements to the Week 24 visit window were < 50 c/mL; denominator was all who remained on treatment through Week 24.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  CVR (n=15, 10, 4, 8, 37) | 4 | 4 | 3 | 4 | 15
  VR-OC (n=11, 10, 4, 7, 32) | 5 | 5 | 2 | 4 | 16

6. Secondary Outcome: Log10 c/mL HIV RNA Changes From Baseline Through Week 48 - Treated Participants
Description: HIV RNA measured as log10 copies per milliliter (c/mL) plasma. HIV RNA values ≥ 1,000 c/mL were considered evidence of infection. A decrease in number of c/mL is an improvement for the participant. HIV RNA was first measured using the ultrasensitive and standard Roche Amplicor PCR, version 1.5, and then the method of measurement was switched to the COBAS AmpliPrep/COBAS TaqMan HIV IVD method. The Baseline visit was within 50 days after the screening visit and was prior to start of study medication (Week 1).
Time Frame: Baseline through Week 48
Population: Treated participants who received at least 1 dose of study drug (EFV) and had an available baseline measurement were analyzed. n=number of participants with available data at both baseline and each specific week.
Measure: Median (Inter-Quartile Range); unit: log10 c/mL
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 13 | 10 | 4 | 7 | 34
log10 c/mL
  Baseline (n=13,10,4,7,34) | 5.88 [5.12 to 5.92] | 5.88 [5.32 to 5.88] | 5.88 [5.38 to 5.88] | 5.50 [4.64 to 5.88] | 5.88 [4.97 to 5.88]
  Week 2 (n=12, 9, 4, 5, 30) | -1.89 (0.270) [-2.60 to -0.93] | -2.26 (0.278) [-2.32 to -1.73] | -2.42 (0.496) [-3.38 to -2.11] | -1.93 (0.277) [-2.49 to -1.85] | -2.11 (0.162) [-2.51 to -1.36]
  Week 4 (n=11, 8, 4, 6, 29) | -2.18 (0.372) [-2.81 to -0.58] | -2.49 (0.308) [-2.86 to -1.86] | -2.86 (0.160) [-3.14 to -2.73] | -3.04 (0.343) [-3.24 to -2.25] | -2.63 (0.195) [-3.06 to -1.69]
  Week 8 (n=11, 10, 3, 7, 31) | -2.73 (0.412) [-3.48 to -0.76] | -2.91 (0.366) [-3.27 to -1.54] | -2.92 (0.070) [-3.12 to -2.90] | -3.27 (0.338) [-4.05 to -2.59] | -2.92 (0.209) [-3.33 to -1.69]
  Week 12 (n=10, 10, 3, 6, 29) | -2.48 (0.541) [-4.00 to -1.33] | -3.19 (0.431) [-3.27 to -1.00] | -4.02 (0.310) [-4.18 to -3.18] | -3.31 (0.362) [-3.87 to -2.95] | -3.14 (0.261) [-3.87 to -1.63]
  Week 16 (n=10, 10, 4, 7, 31) | -2.72 (0.527) [-4.18 to -1.67] | -3.17 (0.496) [-3.55 to -0.44] | -4.11 (0.240) [-4.18 to -3.61] | -3.44 (0.326) [-4.05 to -2.95] | -3.27 (0.253) [-4.05 to -1.94]
  Week 24 (n=10, 9, 3, 7, 29) | -3.46 (0.610) [-4.24 to -1.11] | -3.92 (0.525) [-4.18 to -2.03] | -4.18 (0.585) [-4.18 to -2.43] | -2.95 (0.372) [-4.18 to -2.12] | -3.28 (0.278) [-4.18 to -2.03]
  Week 32 (n=9, 9, 4, 6, 28) | -2.75 (0.547) [-4.08 to -1.67] | -3.28 (0.506) [-4.18 to -1.96] | -3.73 (0.276) [-4.18 to -3.23] | -2.93 (0.461) [-4.18 to -1.69] | -3.27 (0.259) [-4.18 to -1.81]
  Week 40 (n=7, 9, 4 ,6, 26) | -4.01 (0.434) [-4.24 to -1.94] | -4.17 (0.435) [-4.18 to -3.28] | -4.02 (0.236) [-4.18 to -3.52] | -2.93 (0.620) [-4.18 to -0.87] | -3.93 (0.240) [-4.18 to -2.90]
  Week 48 (n=9, 9, 3, 6, 27) | -2.92 (0.551) [-4.18 to -1.67] | -3.27 (0.469) [-4.18 to -1.95] | -3.27 (0.320) [-4.18 to -3.18] | -2.93 (0.622) [-4.18 to -1.69] | -3.18 (0.271) [-4.18 to -1.69]

7. Secondary Outcome: CD4 Cell Count Change From Baseline at Weeks 24 and 48 - Treated Participants
Description: A CD4 cell is an antigenic marker of helper/inducer T cells. These cells were counted during the hematology cell counts performed during a Complete Blood Cell count (CBC) performed by the Central Laboratory. CD4 are measured as number of cells per millimeters to the third power (cells/mm^3). An increase from baseline in the number of CD4 cells is an improvement. The Baseline visit was within 50 days after the screening visit and was prior to start of study medication (Week 1).
Time Frame: Baseline to Weeks 24 and 48
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 10 | 9 | 3 | 6 | 28
cells/mm^3
  Baseline (n=10, 9, 3, 6, 28) | 1518 [829 to 2202] | 1569 [1149 to 2284] | 517 [129 to 558] | 413 [23 to 688] | 1144 [529 to 1930]
  Week 24 (n=6, 7, 3, 6, 22) | 259 (410.8) [-180 to 840] | 82 (330) [-436 to 669] | 31 (818.3) [15 to 2478] | 283 (195.2) [146 to 452] | 177 (185.3) [15 to 669]
  Week 48 (n=7, 8, 2, 5, 22) | -258 (401.5) [-1313 to 606] | 346 (381.8) [-622 to 846] | 971 (956.0) [15 to 1927] | 284 (296.8) [215 to 330] | 196 (220.8) [-258 to 721]

8. Secondary Outcome: Percent of CD4 Cells Change From Baseline at Weeks 24 and 48 - Treated Participants
Description: A CD4 cell is an antigenic marker of helper/inducer T cells. These cells were counted during the hematology cell counts performed during a Complete Blood Cell count (CBC) performed by the Central Laboratory. CD4 are measured as number of cells per millimeter to the third power (cells/mm^3). Percent of CD4 cells is the number of CD4 cells per total number of cells measured*100. An increase in the percent of CD4 cells is an improvement. The Baseline visit was within 50 days after the screening visit and was prior to start of study medication (Week 1).
Time Frame: Baseline to Weeks 24 and 48
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 7 | 9 | 3 | 5 | 24
percentage of CD4 cells
  Baseline (n=7, 9, 3, 5, 24) | 28 [17 to 40] | 26 [25 to 28] | 12 [5 to 20] | 7 [2 to 23] | 24 [14 to 28]
  Week 24 (n=3, 7, 3, 5, 18) | 14 (12.0) [-19 to 19] | 2 (2.8) [0 to 14] | 9 (3.2) [-1 to 9] | 10 (4.2) [9 to 16] | 9 (2.3) [0 to 14]
  Week 48 (n=5, 8, 2, 5, 20) | 5 (4.5) [-2 to 7] | 4 (3.5) [-4 to 11] | 8 (8.9) [-1 to 17] | 11 (2.9) [9 to 12] | 6 (2.1) [-1 to 13]

9. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) Over One Dosing Interval From Time Zero to 24 Hours Post-dose(TAU) at Week 2 - Pharmacokinetic Evaluable Population
Description: Plasma concentrations were obtained using a validated liquid chromatography tandem mass spectrometry method (LC-MS/MS). The lower limit of quantification (LLOQ) for EFV was 10.0 nanograms per milliliter (ng/mL) and the upper limit of quantification (ULOQ) was 8,000 ng/mL. AUC(TAU) was calculated by log- and linear trapezoidal summations. If a concentration was < LLOQ at time TAU, the value of the concentration at time TAU was estimated using the quotient of the last quantifiable concentration and λ. Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the pharmacokinetic parameters summarized using geometric means. AUC(TAU) was measured in micromolars*time (µM•h).
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM•h
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 3 | 10 | 3 | 7
µM•h | 129.5 (98) | 71.4 (49) | 93.8 (68) | 130.8 (98)

10. Primary Outcome: Apparent Oral Clearance (CLT/F) of EFV at Week 2 - Pharmacokinetic Evaluable Population
Description: Plasma concentrations of EFV were obtained using a validated liquid chromatography tandem mass spectrometry method (LC-MS/MS). The lower limit of quantification (LLOQ) for EFV was 10.0 nanograms per milliliter (ng/mL) and the upper limit of quantification (ULOQ) was 8,000 ng/mL. CLT/F was calculated by dividing the dose of EFV by AUC(TAU) of EFV. Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the pharmacokinetic parameters were summarized using geometric means. CLT/F was measured in liters per hour (L/h).
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 3 | 10 | 3 | 7
L/h | 9.54 (63) | 19.69 (85) | 13.16 (58) | 9.11 (73)

11. Primary Outcome: Apparent Oral Clearance Adjusted for Body Weight (CLT/F/kg) of EFV at Week 2 - Pharmacokinetic Evaluable Population
Description: Plasma concentrations of EFV were determined using a validated liquid chromatography tandem mass spectrometry method (LC-MS/MS). The lower limit of quantification (LLOQ) for EFV was 10.0 nanograms per milliliter (ng/mL) and the upper limit of quantification (ULOQ) was 8,000 ng/mL. CLT/F/kg was calculated by dividing CLT/F by body weight in kilograms (kg). Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the pharmacokinetic parameters were summarized using geometric means. CLT/F/kg was measured in liters per hour per kilogram (L/h/kg).
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/kg
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 3 | 10 | 3 | 7
L/h/kg | 2.07 (71) | 2.36 (84) | 1.44 (51) | 0.66 (72)

12. Secondary Outcome: Number of Participants With On-Treatment Adverse Events (AEs), Related Adverse Events, Serious Adverse Events (SAEs), Death, Discontinuation Due to Adverse Events, and CDC Class C AIDS Events
Description: Center for Disease Control and Prevention (CDC) classification of Class C events used to define acquired immunodeficiency syndrome (AIDS): include pneumocystis pneumonia, pneumonia, pulmonary tuberculosis. AE=new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. AE Severity: Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling (Division of AIDs Table, published December 2004). Baseline=within 50 days post screening, prior to start of study drug. 2 categories for death presented (on-treatment and enrolled/not treated).
Time Frame: Baseline to Week 96
Population: All categories except one analyzed treated participants, who received at least 1 dose of study drug (EFV). One category analyzed enrolled participants who were not treated and cannot be assigned to a group.
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  Death (Treated Participants) | 1 | 0 | 1 | 0 | 2
  Deaths (Enrolled Participants, Not treated) | 2 | 0 | 0 | 0 | 2
  SAE (Treated Participants) | 8 | 5 | 4 | 3 | 20
  AE (All Grades,Treated Participants) | 13 | 9 | 4 | 6 | 32
  Grade 2 - 4 AEs (Treated Participants) | 11 | 7 | 4 | 5 | 27
  Grade 3 - 4 AEs (Treated Participants) | 4 | 2 | 3 | 1 | 10
  Related AE (All Grades,Treated Participants) | 8 | 5 | 4 | 4 | 21
  Discontinued due to AE (Treated Participants) | 2 | 0 | 0 | 0 | 2
  CDC Class C AIDS event (Treated Participants) | 1 | 1 | 0 | 0 | 2

13. Secondary Outcome: Number of Participants With Liver Function Test Laboratory Abnormalities - Treated Population
Description: Abnormalities were determined from laboratory measurements analyzed at the central or local laboratory. Division of AIDS Table (DAIDS) for Grading Severity of Adult and Pediatric AEs version (v) Dec 2004. Upper limit of normal (ULN): lower limit of normal (LLN), alanine transaminase (ALT); aspartate aminotransferase (AST); alkaline phosphatase (ALP). ALT Grade (Gr) 1: 1.25 to 2.5*ULN; Gr 2: 2.6 to 5.0*ULN; Gr 3: 5.1 to 10.0*ULN; Gr 4: >10.0*ULN. AST Gr 1: 1.25 to 2.5*ULN; Gr 2: 2.6 to 5.0*ULN; Gr 3: 5.1 to 10.0*ULN; Gr 4: >10.0*ULN. Total bilirubin Gr 1: 1.25 to 1.5*ULN; Gr 2: 1.6 to 2.5*ULN; Gr 3: 2.6 to 5.0*ULN; Gr 4: >5.0*ULN. ALP (U/L) Gr 1: 1.25 to 2.5*ULN, Gr 2: 2.6 to 5.0*ULN, Gr 3: 5.1 to 10.0*ULN, Gr 4: >10.0*ULN. Albumin (low) Gr 1: 3 grams per deciliter (g/dL) to <LLN ; Gr 2: 2.0-2.9 g/dL; Gr 3: < 2 g/dL. Gr 4: Not applicable. Baseline visit was within 50 days after the screening visit and was prior to start of study medication (Week 1).
Time Frame: Baseline to Week 96
Population: Treated participants, who received at least 1 dose of study drug (EFV) were analyzed. n=number of treated participants with available on-treatment data (laboratory measurements).
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  Albumin (n=12, 10, 4, 7, 33) | 0 | 0 | 1 | 0 | 1
  ALP (n=12, 10, 4, 7, 33) | 8 | 2 | 2 | 5 | 17
  ALT (n=12, 10, 4, 7, 33) | 7 | 3 | 2 | 0 | 12
  AST (n=12, 10, 4, 7, 33) | 8 | 1 | 1 | 0 | 10

14. Secondary Outcome: Number of Participants With Lipid and Glucose Laboratory Abnormalities - Treated Participants
Description: Abnormalities were determined from measurements analyzed at central or local laboratory. DAIDS Grading Severity of Adult and Pediatric AEs v Dec 2004. Total Cholesterol (fasting) Gr 1: 170 - 199 mg/dL; Gr 2: 200 - 300 mg/dL; Gr 3 >300 mg/dL; Gr 4 Not Applicable(NA). LDL cholesterol, fasting: Gr 1: 110-129 mg/dL; Gr 2: 130-189 mg/dL; Gr 3 >=190 mg/dL; Gr 4 NA. Triglycerides, fasting: Gr 1: NA; Gr 2 500-750 mg/dL; Gr 3: 751-1,200 mg/dL; Gr 4: >1,200 mg/dL. Glucose, serum, high, fasting and (non-fasting): Gr 1: 110 - 125 (116-160) mg/dL; Gr 2: 126-250 (161- 250) mg/dL; Gr 3: 251-500 (251-500) mg/dL; Gr 4: >500 (> 500) mg/dL. Glucose, serum, low, >=1 month of age (<1 month): Gr 1: 55-64 (50-54) mg/dL; Gr 2: 40-54 (40-49) mg/dL; Gr 3: 30-39 (30-39) mg/dL; Gr 4: <30 (<30) mg/dL. Baseline: within 50 days after the screening visit and was prior to start of study medication (Week 1). Only those in 4th arm were old enough to fast prior to testing; other arms did not have fasting samples taken.
Time Frame: Baseline to Week 96
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  Total Cholesterol (n=9,10,4,0,23) | 2 | 4 | 1 | NA — only fasting samples taken | 7
  Total Cholesterol Fasting (n=0,0,0,7,7) | NA — too young to fast, samples not taken | NA — too young to fast, samples not taken | NA — too young to fast, samples not taken | 1 | 1
  Glucose High (n=11,10,3,0,24) | 1 | 0 | 0 | NA — only fasting samples taken | 1
  Glucose Low (n=11,10,3,0,24) | 2 | 1 | 0 | NA — only fasting samples taken | 3
  Glucose High Fasting (n=0,0,0,7,7) | NA — too young to fast, samples not taken | NA — too young to fast, samples not taken | NA — too young to fast, samples not taken | 1 | 1
  LDL cholesterol (n=9,10,4,0,23) | 0 | 4 | 0 | NA — only fasting samples taken | 4
  LDL cholesterol fasting (n=0,0,0,7,7) | NA — too young to fast, samples not taken | NA — too young to fast, samples not taken | NA — too young to fast, samples not taken | 1 | 1

15. Secondary Outcome: Number of Participants With Serum Chemistry Abnormalities - Treated Participants
Description: Central/local laboratory. DAIDS v 2004. Bicarbonate, low: Gr 1: 16 milliequivalents per liter (mEq/L) - < LLN; Gr 2: 11.0-15.9 mEq/L; Gr 3: 8.0-10.9 mEq/L; Gr 4: <8.0 mEq/L; calcium, high Gr 1: 10.6-11.5 mg/dL; Gr 2: 11.6-12.5 mg/dL; Gr 3 12.6-13.5 mg/dL; Gr 4: >13.5 mg/dL; calcium, low Gr1: 7.8-8.4 mg/dL; Gr2: 7.0-7.7 mg/dL; Gr3: 6.1-6.9 mg/dL; Gr 4: <6.1 mg/dL; creatinine Gr1: 1.1-1.3*ULN; Gr 2: 1.4-1.8*ULN; Gr 3: 1.9-3.4*ULN; Gr 4: >=3.5*ULN; lipase Gr 1: 1.1-1.5*ULN; Gr 2: 1.6-3.0*ULN; Gr 3: 3.1-5.0*ULN; Gr 4: >5.0*ULN; potassium high (low) Gr 1: 5.6-6.0 (3.0-3.4) mEq/L; Gr 2: 6.1-6.5 (2.5-2.9) mEq/L; Gr 3: 6.6-7.0 (2.0-2.4) mEq/L; Gr 4: >7.0 (<2.0) mEq/L; sodium, high (low) Gr 1: 146-150 (130-135) mEq/L; Gr 2: 151-154 (125-129) mEq/L; Gr 3: 155-159 (121-124) mEq/L; Gr 4: >=160 (<=120) mEq/L; uric acid Gr 1: 7.5-10.0 mg/dL; Gr 2: 10.1-12.0 mg/dL; Gr 3: 12.1-15.0 mg/dL; Gr 4: >15.0 mg/dL. Baseline within 50 days post screening, prior to start of study medication.
Time Frame: Baseline to Week 96
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  Bicarbonate, low (n=12, 10, 4, 7, 33) | 10 | 9 | 4 | 5 | 28
  Sodium, low (n=12, 10, 4, 7, 33) | 5 | 4 | 2 | 4 | 15
  Sodium High (n=12, 10, 4, 7, 33) | 1 | 1 | 0 | 1 | 3
  Uric Acid (n=12, 10, 4, 7, 33) | 0 | 1 | 1 | 0 | 2
  Calcium High (n= 12, 10, 4, 7, 33) | 0 | 2 | 0 | 1 | 3
  Calcium Low (n= 12, 10, 4, 7, 33) | 0 | 4 | 1 | 1 | 6
  Potassium High (n= 12, 10, 4, 7, 33) | 5 | 4 | 0 | 0 | 9
  Potassium Low (n= 12, 10, 4, 7, 33) | 1 | 0 | 1 | 1 | 3
  Lipase Total (n= 12, 10, 4, 7, 33) | 1 | 0 | 0 | 2 | 3

16. Secondary Outcome: Number of Participants With Hematologic Abnormalities - Treated Participants
Description: Abnormalities were determined from laboratory measurements analyzed at the central or local laboratory. DAIDS DAIDS Grading Severity of Adult and Pediatric AEs v Dec 2004. Hemoglobin Gr 1: 8.5-10.0 g/dL; Gr 2: 7.5-8.4 g/dL; Gr 3: 6.50-7.4 g/dL; Gr 4: <6.5 g/dL; Platelets, decreased: Gr 1: 100.000-124.999*10^9/L; Gr 2: 50.000-99.999*10^9/L; Gr 3: 25.000-49.999*10^9/L; Gr 4: <25.000*10^9/L; White blood cell count (WBC) decreased Gr 1: 2.000-2.500*10^9/L; Gr 2: 1.500-1.999*10^9/L; Gr 3: 1.000-1.499*10^9/L; Gr 4: <1.000*10^9/L. Baseline visit was within 50 days post screening and was prior to start of study drug (Week 1).
Time Frame: Baseline to Week 96
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  Hemoglobin (n=11, 10, 4, 7, 32) | 4 | 5 | 2 | 1 | 12
  Platelet (n=11, 10, 4, 7, 32) | 1 | 1 | 0 | 0 | 2
  Neutrophils (n=11, 10, 4, 7, 32) | 7 | 2 | 0 | 1 | 10

17. Secondary Outcome: Number of Treated Participants With Resistance Associated Genotypic and Phenotypic Changes in Viruses - Participants With Virologic Failure, Lack of Suppression or Viral Load Rebound
Description: At baseline, treatment-naïve screened by genotype; treatment-experienced screened by genotype and phenotype. Genotypic resistance: presence of substitutions in reverse transcriptase (RT) gene and/or presence of mutations that confer resistance to nucleoside reverse transcriptase inhibitor class. Phenotype resistance: FTC: > 3.1* the 50% inhibitory concentration (IC50) of the control strain; EFV: > 3.3* IC50 ; ddI: > 2.6*IC50. Virologic failure: <1 log10 decrease in HIV RNA from Week 16 on; confirmatory HIV RNA within 14-35 days; HIV RNA > 10,000 c/mL with prior value < 400 c/mL; confirmatory HIV RNA 14-35 days. Monogram Biosciences Phenosense™ assay ( EFV and FTC: biologic cutoffs=3 and 3.5, respectively; ddI: clinical cutoff: lower limit=1.39; upper limit = 2.2.); VircoTYPE™ HIV-1 v 4.3.01( EFV, FTC: biologic cutoffs=3.3 and 3.1, respectively;ddI: clinical cutoff: lower limit = 0.9; upper limit = 2.6. No genotypic/phenotypic changes in presence of virologic failure=no resistance.
Time Frame: Baseline to Week 48
Population: Participants who met the definition of virologic failure per protocol (PP): n=6 ; in addition, those who rebounded on treatment with plasma HIV RNA > 10,000 c/mL but samples were not obtained within specified 35 day limit were included (not PP): n=5; participants with virologic failure and with samples available for analysis of virus changes:n=11.
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 4 | 5 | 1 | 1 | 11
participants
  Lack of suppression with Changes (PP) | 2 | 1 | 0 | 0 | 3
  Viral Load Rebound with Changes(PP) | 1 | 1 | 0 | 0 | 2
  Viral Failure with Changes (outside 35 day limit) | 0 | 3 | 1 | 1 | 5

18. Secondary Outcome: Number of Participants With Acquisition of Resistance to EFV Categorized by AUC Relationship - Evaluable Pharmacokinetic Population
Description: PK parameters were evaluated 2 weeks post start of dosing. Based on observed AUC, measured in micromoles (μM)*h, dosing was increased, remained the same, or decreased at next visit to achieve the desired AUC (110-380 μM*h). Number of participants who became resistant was categorized by those who required additional dosing after Week 2 (AUC<110 μM*h) and those who did not. AUC: derived from plasma concentration of EFV versus time. Plasma concentrations for determination of AUC were obtained using a validated LC-MS/MS method. LLOQ for EFV = 10.0 ng/mL and ULOQ = 8,000 ng/mL. AUC calculated by log- and linear trapezoidal summations. Genotypic resistance=presence of substitutions in the RT gene and/or presence of mutations that confer resistance to entire nucleoside reverse transcriptase inhibitor class. Phenotypic resistance=EFV: > 3.3* IC50 of control strain. Assays: Monogram Biosciences Phenosense™ GT (EFV biologic cutoff=3) and VircoTYPE™ HIV-1 v 4.3.01( EFV biologic cutoff=3.3).
Time Frame: Baseline to Week 48
Population: All participants who received at least one dose of study drug (EFV) and had adequate pharmacokinetic (PK) profiles at Week 2 were analyzed. n=number of participants with AUC<110 µM•h and number of participants with AUC>=110 µM•h.
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 12 | 10 | 4 | 7 | 33
participants
  Resistant; AUC<110 µM•h(n=2,7,2,3,14) | 1 | 3 | 1 | 1 | 6
  Resistant; AUC>=110 µM•h(n=10,3,2,4,19) | 2 | 2 | 0 | 0 | 4

19. Secondary Outcome: Cmax and Cmin of Didanosine (ddI) at Week 2 - Pharmacokinetic Evaluable Population
Description: Cmax and Cmin were derived from plasma concentration versus time. Plasma concentrations for ddI were determined using a validated LC/MS/MS assay. All reportable Cmin values were <LLOQ in all age groups except >=6 months to < 2 years (Group 2); LLOQ/2 was imputed for those summary statistics;in Group 2, 9 of 10 Cmin values were <LLOQ; LLOQ/2 was imputed for those samples for summary statistics. The lower limit of quantification (LLOQ) for ddI was 2.50 nanograms per milliliter (ng/mL). Cmax and Cmin were recorded directly from experimental observations. Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the pharmacokinetic parameters were summarized using geometric means. Cmax and Cmin were measured in ng/mL.
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- EFV+ddI+FTC in Infants >=3 Months to < 6 Months; EFV+ddI+FTC in Infants >=6 Months to < 2 Years; EFV+ddI+FTC in Children >= 2 Years to < 3 Years; EFV+ddI+FTC in Children >= 3 Years to <= 6 Years: EFV (efavirenz) was administered in accordance with weight-based dosing nomograms and included one of the following preparations in a once a day (QD) dose: EFV capsules (50 and 200 mg) contents mixed with formula or a small amount of food vehicle (eg, yogurt, applesauce, or grape jelly), or oral solution (30 mg/mL); participants unable to meet the desired exposures using the oral solution, or those not able to tolerate the oral solution, used the capsule contents sprinkled on food. In addition, the following 2 drugs were administered: ddI (didanosine) (Pediatric Powder for Oral Solution or capsules of enteric-coated beads): 240 mg/m^2 QD; maximum daily dose of 400 mg and FTC (emtricitabine) (solution or tablets) 6 mg/kg QD; maximum daily dose of 240 mg.
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 12 | 10 | 4 | 6
ng/mL
  Cmax (n=12, 10, 4, 6) | 850 (48) | 1193 (39) | 356 (69) | 376 (93)
  Cmin (n=4, 10, 4, 3) | 1.25 (0) | 1.54 (132) | 1.25 (0) | 1.25 (0)

20. Secondary Outcome: AUC (TAU) of Didanosine (ddI) at Week 2 - Pharmacokinetic Evaluable Population
Description: Plasma concentrations were obtained using a validated LC-MS/MS at Week 2. The lower limit of quantification (LLOQ) for ddI was 2.50 nanograms per milliliter (ng/mL). AUC(TAU) was calculated by log- and linear trapezoidal summations. If a concentration was < LLOQ at time TAU, the value of the concentration at time TAU was estimated using the quotient of the last quantifiable concentration and λ. Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the pharmacokinetic parameters summarized using geometric means. AUC(TAU) was measured in nanograms*time per milliliter (ng•h/mL).
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 4 | 10 | 4 | 4
ng•h/mL | 1445 (76) | 2848 (53) | 1038 (54) | 1000 (41)

21. Secondary Outcome: CLT/F of Didanosine (ddI) at Week 2 - Pharmacokinetic Evaluable Population
Description: Plasma concentrations for ddI were determined using a validated LC/MS/MS assay. The LLOQ for ddI was 2.50 nanograms per milliliter (ng/mL). CLT/F was calculated by dividing the dose of ddI by AUC(TAU) of ddI. Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the pharmacokinetic parameters were summarized using geometric means. CLT/F was measured in liters per hour (L/h).
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 4 | 10 | 4 | 4
L/h | 40.7 (110) | 35.6 (42) | 113.9 (111) | 143.0 (53)

22. Secondary Outcome: CLT/F/kg of Didanosine (ddI) at Week 2 - Pharmacokinetic Evaluable Population
Description: Plasma concentrations for ddI were determined using a validated LC/MS/MS assay. The LLOQ for ddI was 2.50 nanograms per milliliter (ng/mL). CLT/F/kg was calculated by dividing CLT/F by body weight in kilograms (kg). Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the pharmacokinetic parameters were summarized using geometric means. CLT/F/kg was measured in liters per hour per kilogram (L/h/kg).
Time Frame: Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/kg
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 4 | 10 | 4 | 4
L/h/kg | 7.88 (85) | 4.26 (30) | 11.36 (116) | 10.34 (70)

23. Secondary Outcome: Terminal Phase Elimination Half-life (T-HALF) in Didanosine (ddI) at Week 2 - Pharmacokinetic Evaluable Population
Description: Plasma concentrations for ddI were determined using a validated LC/MS/MS assay. The LLOQ for ddI was 2.50 nanograms per milliliter (ng/mL). Blood samples were collected before study drug administration and at 0.5, 1, 3, 5, 8, and 24 hours after study drug administration from an indwelling catheter or by direct venipuncture and the T-HALF was summarized using a mean. Terminal elimination plasma half-life=ln2 divided by K where K is the absolute value of the slope of the terminal phase of the plasma profile as determined by log-linear regression of at least three data points. T-HALF was measured in hours (h).
Time Frame: Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years
Number analyzed (Participants) | 3 | 10 | 4 | 4
h | 0.92 (0.1374) | 1.41 (0.859) | 1.73 (1.007) | 1.14 (0.214)

24. Secondary Outcome: The Number of Participants With Plasma HIV RNA Levels < 400 c/mL at Weeks 60, 72, 84 and 96 (Observed Cases) - All Treated Participants
Description: Virologic Response - Observed Cases (VR-OC): participants were responders at a specific week according to a single on-treatment HIV RNA < 400 c/mL closest to the planned visit and within the predefined visit window; those on treatment and missing their specific week measurement were responders only if previous and subsequent measurements to that week visit window were < 400 c/mL; denominator was all who remained on treatment through the specific week.
Time Frame: Weeks 60, 72, 84, and 96
Population: Treated participants, who received at least 1 dose of study drug (EFV) were analyzed. n=number of treated participants with available on-treatment data at each specific week.
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  Week 60 (n=7, 8, 3, 4, 22) | 7 | 6 | 2 | 4 | 19
  Week 72 (n=7, 7, 2, 4, 20) | 7 | 5 | 1 | 4 | 17
  Week 84 (n=7, 7, 2, 4, 20) | 7 | 5 | 1 | 4 | 17
  Week 96 (n=7, 6, 2, 4, 19) | 7 | 5 | 1 | 4 | 17

25. Secondary Outcome: The Number of Participants With Plasma HIV RNA Levels < 50 c/mL at Weeks 60, 72, 84 and 96 (Observed Cases) - All Treated Participants
Description: Virologic Response - Observed Cases (VR-OC): participants were responders at a specific week according to a single on-treatment HIV RNA < 50 c/mL closest to the planned visit and within the predefined visit window; those on treatment and missing their specific week measurement were responders only if previous and subsequent measurements to that week visit window were < 50 c/mL; denominator was all who remained on treatment through the specific week.
Time Frame: Weeks 60, 72, 84, and 96
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 15 | 10 | 4 | 8 | 37
participants
  Week 60 (n=7, 8, 3, 4, 22) | 4 | 5 | 2 | 3 | 14
  Week 72 (n=7, 7, 2, 4, 20) | 7 | 5 | 1 | 4 | 17
  Week 84 (n=7, 7, 2, 4, 20) | 7 | 5 | 1 | 3 | 16
  Week 96 (n=7, 6, 2, 4, 19) | 6 | 5 | 0 | 4 | 15

26. Secondary Outcome: Log10 c/mL HIV RNA Changes From Baseline at Weeks 60, 72, 84 and 96 - Treated Participants
Description: as for outcome 6
Time Frame: Baseline through Weeks 60, 72, 84, and 96
Population: Treated participants who received at least 1 dose of study drug (EFV) were analyzed. n=number of participants with available data at both baseline and each specific week on treatment.
Measure: Median (Inter-Quartile Range); unit: log10 c/mL
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 13 | 10 | 4 | 7 | 34
log10 c/mL
  Baseline (n=13,10,4,7,34) | 5.88 [5.12 to 5.92] | 5.88 [5.32 to 5.88] | 5.88 [5.38 to 5.88] | 5.50 [4.64 to 5.88] | 5.88 [4.97 to 5.88]
  Week 60 (n=7, 8, 3, 4, 22) | -3.92 (0.458) [-418 to -1.94] | -3.44 (0.539) [-4.18 to -1.46] | -3.26 (0.322) [-4.18 to -3.18] | -3.48 (0.575) [-4.10 to -2.32] | -3.50 (0.259) [-4.18 to -1.94]
  Week 72 (n=7, 6, 1, 3, 17) | -4.08 (0.438) [-4.24 to -1.94] | -2.75 (0.603) [-418 to -1.83] | -3.20 (NA) [-3.20 to -3.20] | -4.18 (0.410) [-4.18 to -2.95] | -3.45 (0.290) [-4.18 to -2.21]
  Week 84 (n=7, 7, 2, 4, 20) | -4.08 (0.438) [-4.24 to -1.94] | -3.28 (0.563) [-4.18 to -1.54] | -2.18 (1.022) [-3.20 to -1.16] | -3.51 (0.583) [-4.13 to 02.32] | -3.37 (0.283) [-4.18 to -1.81]
  Week 96 (n=7, 6, 2, 4, 19) | -3.82 (0.423) [-4.18 to -1.94] | -3.73 (0.686) [-4.18 to -1.19] | -2.15 (0.848) [-2.99 to -1.30] | -3.57 (0.597) [-4.18 to -2.32] | -3.45 (0.296) [-4.18 to -1.69]

27. Secondary Outcome: CD4 Cell Count Change From Baseline at Weeks 60, 72, 84, and 96 - Treated Participants
Description: as for outcome 7
Time Frame: Baseline to Weeks 60, 72, 84, and 96
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 10 | 9 | 3 | 6 | 28
cells/mm^3
  Baseline (n=10,9,3,6,28) | 1518 [829 to 2202] | 1569 [1149 to 2284] | 517 [129 to 558] | 413 [23 to 688] | 1144 [529 to 1930]
  Week 60 (n=6, 6, 2,3,17) | -870 [-1331 to -315] | -914 [-1509 to 725] | 580 [-11 to 1171] | 676 [506 to 887] | -315 [-1331 to 676]
  Week 72 (n=5, 7, 1, 3, 16) | -1178 [-1422 to -588] | 234 [-1540 to 624] | -50 [-50 to -50] | 620 [619 to 811] | 92 [-1300 to 620]
  Week 84 (n=6, 7, 1, 3, 17) | -937 [-1331 to -155] | 59 [-1416 to 316] | 101 [101 to 101] | 497 [339 to 722] | 59 [-1304 to 334]
  Week 96 (n=6, 6, 1, 3, 16) | -834 [-1437 to -176] | -43 [-1291 to 222] | 402 [402 to 402] | 744 [295 to 1243] | -40 [-1185 to 314]

28. Secondary Outcome: Percent of CD4 Cells Change From Baseline at Weeks 60, 72, 84, and 96 - Treated Participants
Description: as for outcome 8
Time Frame: Baseline to Weeks 60, 72, 84, and 96
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | EFV+ddI+FTC in Infants >=3 Months to < 6 Months | EFV+ddI+FTC in Infants >=6 Months to < 2 Years | EFV+ddI+FTC in Children >= 2 Years to < 3 Years | EFV+ddI+FTC in Children >= 3 Years to <= 6 Years | EFV+ddI+FTC in All Participants
Number analyzed (Participants) | 7 | 9 | 3 | 5 | 24
percentage of CD4 cells
  Baseline (n=7,9,3,5,24) | 28 [17 to 40] | 26 [25 to 28] | 12 [5 to 20] | 7 [2 to 23] | 24 [14 to 28]
  Week 60 (n=3,6,2,3,14) | 10 [-9 to 13] | 3 [-5 to 5] | 7 [-1 to 15] | 13 [9 to 26] | 7 [-1 to 13]
  Week 72 (n=2,7,1,3,13) | -14 [-17 to -10] | 1 [-5 to 13] | -1 [-1 to -1] | 12 [11 to 26] | 1 [-5 to 12]
  Week 84 (n=3,7,1,3,14) | -3 [-22 to 21] | 8 [0 to 11] | 2 [2 to 2] | 12 [5 to 34] | 7 [0 to 12]
  Week 96 (n=3,6,1,3,13) | -2 [-19 to 6] | 7 [3 to 10] | 15 [15 to 15] | 14 [14 to 28] | 7 [3 to 14]

ADVERSE EVENTS:
Time Frame: 96 Weeks (Last patient, last visit).
Description: Participants who received at least one dose of study drug.
Arm/Group | EFV+ddI+FTC in All Participants
Serious Adverse Events (participants affected / at risk) | 20/37
Other Adverse Events (participants affected / at risk) | 30/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EFV+ddI+FTC in All Participants (N=37)
Eczema (Skin and subcutaneous tissue disorders) | 1
Oral herpes (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Epilepsy (Nervous system disorders) | 1
Appendicitis perforated (Infections and infestations) | 1
Bovine tuberculosis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Varicella (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 1
Viral rash (Infections and infestations) | 1
Febrile convulsion (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 8
Gastroenteritis (Infections and infestations) | 3
Mass (General disorders) | 1
Otitis media (Infections and infestations) | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Impetigo (Infections and infestations) | 1
Lymph node tuberculosis (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Oral candidiasis (Infections and infestations) | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EFV+ddI+FTC in All Participants (N=37)
Abdominal pain (Gastrointestinal disorders) | 2
Acarodermatitis (Infections and infestations) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 4
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2
Papule (Skin and subcutaneous tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Bronchitis (Infections and infestations) | 5
Head injury (Injury, poisoning and procedural complications) | 2
Lymph node palpable (Investigations) | 2
Nasopharyngitis (Infections and infestations) | 13
Nausea (Gastrointestinal disorders) | 2
Pharyngotonsillitis (Infections and infestations) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Prurigo (Skin and subcutaneous tissue disorders) | 2
Pyrexia (General disorders) | 9
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Viral rhinitis (Infections and infestations) | 2
Candida nappy rash (Infections and infestations) | 5
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5
Dermatosis (Skin and subcutaneous tissue disorders) | 2
Herpes zoster (Infections and infestations) | 2
Mastoiditis (Infections and infestations) | 2
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2
Otitis media acute (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 2
Steatorrhoea (Gastrointestinal disorders) | 3
Varicella (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 3
Dental caries (Gastrointestinal disorders) | 2
Influenza (Infections and infestations) | 6
Rhinitis (Infections and infestations) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 4
Tonsillitis (Infections and infestations) | 2
Blood alkaline phosphatase increased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 2
Pneumonia (Infections and infestations) | 4
Diarrhoea (Gastrointestinal disorders) | 19
Gastroenteritis (Infections and infestations) | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Otitis media (Infections and infestations) | 7
Stomatitis (Gastrointestinal disorders) | 2
Conjunctivitis (Eye disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Ear infection (Infections and infestations) | 2
Impetigo (Infections and infestations) | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 3
Otitis media chronic (Infections and infestations) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Oral candidiasis (Infections and infestations) | 3
Otitis externa (Infections and infestations) | 2
Product taste abnormal (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.